CLINICAL TRIAL: NCT00876018
Title: A Double Blind Randomized Controlled Trial in School Going Children, to Evaluate the Impact of a Multiple Micronutrient Fortified Nutritional Powder on Physical Performance Measures
Brief Title: Nutrition, Physical Performance & Fitness in Indian School Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IND 001/2008
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Physical Fitness; Nutritional Status
Keywords: physical performance; micronutrients; physical fitness; healthy children
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- No intervention (No Intervention): No intervention
- Nutritional supplement (Experimental): Fortified nutritional powder
  Interventions: Other: Nutritional supplement
- Placebo (Placebo Comparator): Un-fortified nutritional powder
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Nutritional supplement — Fortified nutritional powder
  Arms: Nutritional supplement
Other: Placebo — Un-fortified nutritional powder
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of nutritional supplement on physical performance measures of apparently healthy school going children in India.

DETAILED DESCRIPTION:
Nutritional status may be important in achieving optimal physical performance. There is evidence of significant improvements in physical fitness, aerobic capacity and anaerobic threshold of children and adolescents with nutritional intervention, albeit in children with initial sub-optimal nutritional status. This may be of particular relevance in developing countries like India, where there is limited data on physical fitness and a wide-spread prevalence of concurrent micronutrient deficiencies even in apparently normal school age children. The present study therefore, is designed to assess the effect of a nutritional supplement on the physical performance measures of school going children. This is a randomized, double blind placebo-controlled study of three treatment groups (1 test, 1 positive control (placebo) and 1 'no intervention') conducted in equal numbers of male or female children [ages 7-11] attending day schools in Bangalore. Subjects in the intervention (test and positive control) groups will receive study treatments (fortified or un-fortified nutritional powder) once a day for 4 months. The treatments will be administered under supervision on all school working days; for the weekend and other holidays, sachets will be provided for home consumption. At baseline and 4months, physical performance tests will be administered and blood sample drawn to assess nutritional status. Other selected outcome measures such as nutrition status and muscle strength/ endurance will also be assessed. It is hypothesized that after 4 months of intervention, children consuming fortified nutritional powder will have statistically significant improvements in physical performance/ fitness measures as compared to the two control groups.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls between ages 7-10.5 years
* Z score of height for age and weight for age of 0 to < -3
* Good general health at screening
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Written informed consent from the parents/ guardians and writtent assent by the study participant

Exclusion Criteria:

* Severe anemia (Hb<8 g% )
* Cardiovascular disease on clinical examination or history
* Any underlying respiratory disease with impairment of lung function
* Physical disability Children consuming nutritional supplements (tonics, syrups, tablets or chews) and/ or health food drinks on a regular basis
* Recent history [3mo] of serious infections, injuries and/ or surgeries
* Participation in any nutritional study in the last 1 year
* Indication that they are likely to move within the period of study intervention
* Any known food allergies like peanut allergy, gluten allergy
* Family members of an employee of the Sponsor or the study site.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2008-07-07 (Actual); Primary Completion 2008-12-19 (Actual); Study Completion 2008-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangalore, Karnataka, India

REFERENCES:
- [Derived] Desai IK, Kurpad AV, Chomitz VR, Thomas T. Aerobic fitness, micronutrient status, and academic achievement in Indian school-aged children. PLoS One. 2015 Mar 25;10(3):e0122487. doi: 10.1371/journal.pone.0122487. eCollection 2015. PMID 25806824
- [Derived] Vaz M, Pauline M, Unni US, Parikh P, Thomas T, Bharathi AV, Avadhany S, Muthayya S, Mehra R, Kurpad AV. Micronutrient supplementation improves physical performance measures in Asian Indian school-age children. J Nutr. 2011 Nov;141(11):2017-23. doi: 10.3945/jn.110.135012. Epub 2011 Sep 14. PMID 21918063

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three schools of Karnataka at a clinical site in Karnataka.
Pre-assignment Details: A total of 379 participants were screened. Out of which 300 participants were randomized.
Groups:
- Experimental Group (Fortified Nutritional Supplement): Participants were administered with fortified choco-malt beverage powder (including 19 key vitamins and minerals) as single serves of 40 gram (g) in 100 milliliter (mL) water. Administration was done once a day for 4 months under study personnel supervision on all school working days (6 days per week) and for self-consumption on weekends and/ or holidays.
- Control Group A (Un-fortified Nutritional Powder): Participants were administered with unfortified choco-malt beverage powder (energy equivalent of fortified choco-malt powder in experimental group) as single serves of 40g in 100mL water. Administration was done once a day for 4 months under study personnel supervision on all school working days (6 days per week) and for self-consumption on weekends and/ or holidays.
- Control Group B (No Intervention): Participants were not administered with any intervention.
Period: Overall Study
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Un-fortified Nutritional Powder) | Control Group B (No Intervention)
Started | 100 | 100 | 100
Completed | 95 | 95 | 97
Not Completed | 5 | 5 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrew Consent due to Adverse Event | 5 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group (Fortified Nutritional Supplement): Participants were administered with fortified choco-malt beverage powder as single serves of 40g in 100mL water. Administration was done once a day for 4 months under study personnel supervision on all school working days (6 days per week) and for self-consumption on weekends and/ or holidays.
- Control Group A (Unfortified Nutritional Powder): Participants were administered with unfortified choco-malt beverage powder (energy equivalent of fortified choco-malt powder in experimental group). Administration was done once a day for 4 months under study personnel supervision on all school working days (6 days per week) and for self-consumption on weekends and/ or holidays.
- Total: Total of all reporting groups
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention) | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.26 (1.02) | 8.18 (1.01) | 8.29 (1.04) | 8.24 (1.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 50 | 150
  Male | 50 | 50 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maximal Aerobic Capacity (VO2max)- 12 Inch Step Test After 4 Months
Description: Maximal aerobic capacity (VO2max) is defined as the maximum rate of oxygen consumption, measured during incremental exercise. VO2max was measured with the help of an externally placed 12-inch step test to assess the aerobic fitness/cardio-respiratory endurance of the study participants. In this test, participants were asked to step at 22 steps a minute for 3 minutes. The pulse rate was recorded manually, within 15sec of stopping the test. VO2max was calculated as (VO2 x HRmax) divided by HR observed, where HRmax = 220-Age in years. HRmax= maximum heart rate. VO2 is equal to (0.2 x Stepping Rate) + (2.4 x Step height x Stepping Rate) + 3.5 mL/kg/min. mL/kg/min.= milliliter per kilogram per minute.
Time Frame: Baseline, after 4 months
Population: Analysis for this outcome was performed on all randomized population. Number of participants analyzed is the number of participants from the randomized population evaluated at specific time points for respective treatment arm.
Measure: Mean (Standard Deviation); unit: mL/kg/min.
Groups:
- Experimental Group (Fortified Nutritional Supplement): Participants were administered with fortified choco-malt beverage powder (including 19 key vitamins and minerals) as single serves of 40g in 100mL water. Administration was done once a day for 4 months under study personnel supervision on all school working days (6 days per week) and for self-consumption on weekends and/ or holidays.
- Control Group A (Unfortified Nutritional Powder): Participants were administered with unfortified choco-malt beverage powder (energy equivalent of fortified choco-malt powder in experimental group) as single serves of 40g in 100mL water. Administration was done once a day for 4 months under study personnel supervision on all school working days (6 days per week) and for self-consumption on weekends and/ or holidays.
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
mL/kg/min.
  At Baseline: number analyzed (Participants) | 99 | 100 | 99
  At Baseline | 36.8 (5.3) | 37.9 (5.6) | 37.0 (5.3)
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 38.9 (5.6) | 37.6 (5.3) | 37.8 (5.3)
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Change from baseline after 4 months | 2.00 (6.03) | -0.25 (6.23) | 0.7 (5.87)
Statistical Analysis 1: Comparison: Experimental Group (Fortified Nutritional Supplement) vs Control Group A (Unfortified Nutritional Powder); Test type: Other; p = 0.004, Mann Whitney U test
Statistical Analysis 2: Comparison: Experimental Group (Fortified Nutritional Supplement) vs Control Group B (No Intervention); Test type: Other; p = 0.147, Mann Whitney U test

2. Primary Outcome: Change From Baseline in Aerobic Capacity-shuttle Test (VO2peak) After 4 Months
Description: Aerobic capacity(VO2peak) is defined as maximum rate of oxygen consumption attained on a particular exercise test. VO2peak was measured by 20m shuttle run test to assess aerobic & whole body endurance. In this test, participants were asked to move around one cone to another placed at 19m distance, reversing direction & in accordance with a pace dictated by sound signal, that got progressively faster at one minute intervals. The initial pace was set at 4.0 km/hr & with subsequent increases of 0.5 km/hr every subsequent minute. This test was conducted in groups (of at least 3 children per group). The shuttle was stopped when either the participant chose to stop because of exhaustion or when participant was > 1m away from cone at 2 consecutive paced signals. The number of shuttles at stoppage was noted. VO2peak was calculated as 31.025 + (3.325 x speed) - (3.248 x age). Speed is speed attained in previous level of shuttle, computed as speed (km/hr) = v + 0.5 x n/60; and age is in years.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: km/hr*years
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
km/hr*years
  At Baseline | 31.6 (4.3) | 32.8 (4.1) | 32.4 (4.2)
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 39.1 (4.3) | 38.6 (3.7) | 38.2 (4.1)
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Change from baseline after 4 months | 7.52 (3.51) | 5.74 (6.02) | 5.80 (3.56)
Statistical Analysis 1: Comparison: Experimental Group (Fortified Nutritional Supplement) vs Control Group A (Unfortified Nutritional Powder); Test type: Other; p = 0.002, Mann Whitney U test
Statistical Analysis 2: Comparison: Experimental Group (Fortified Nutritional Supplement) vs Control Group B (No Intervention); Test type: Other; p = 0.003, Mann Whitney U test

3. Primary Outcome: Change From Baseline in Time Taken for 40 Meter (m) Sprint After 4 Months
Description: A 40m sprint was used to assess speed with time taken to complete the sprint being recorded manually using a digital stopwatch. The moment any part of the designated participant's body reached the marker level, the corresponding examiner stopped their watches and recorded the time for the sprint.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds (Sec)
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
seconds (Sec)
  At Baseline | 9.0 (1.3) | 8.9 (1.0) | 8.9 (1.0)
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 8.6 (1.1) | 8.9 (1.0) | 8.639 (1.0)
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Change from baseline after 4 months | -0.34 (0.99) | -0.05 (0.93) | -0.26 (1.0)
Statistical Analysis 1: Comparison: Experimental Group (Fortified Nutritional Supplement) vs Control Group A (Unfortified Nutritional Powder); Test type: Other; p = 0.153, Mann Whitney U test
Statistical Analysis 2: Comparison: Experimental Group (Fortified Nutritional Supplement) vs Control Group B (No Intervention); Test type: Other; p = 0.903, Mann Whitney U test

4. Primary Outcome: Change From Baseline in Visual Reaction Time After 4 Months
Description: Visual reaction time was assessed using a customized computer based programme. Participant was provided with a periodic random test visual stimulus among many other 'non test' stimuli. Participant was required to tap the space bar of the computer as fast as possible on the appearance of the test visual stimulus. Three test visual cues were provided at each sitting to allow for training effects. The shortest visual reaction time of the three visual cues was used in analyses.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
milliseconds (msec)
  At Baseline | 958 (217) | 932 (189) | 939 (210)
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 863 (144) | 884 (122) | 864 (157)
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Change from baseline after 4 months | -94 (227) | -46 (180) | -72 (249)
Statistical Analysis 1: Comparison: Experimental Group (Fortified Nutritional Supplement) vs Control Group A (Unfortified Nutritional Powder); Test type: Other; p = 0.143, Mann Whitney U test
Statistical Analysis 2: Comparison: Experimental Group (Fortified Nutritional Supplement) vs Control Group B (No Intervention); Test type: Other; p = 0.678, Mann Whitney U test

5. Secondary Outcome: Change From Baseline in Maximal Handgrip Strength for Dominant and Non-dominant Hand After 4 Months
Description: Maximal handgrip strength was measured using a Jamar handgrip dynamometer in dominant and non-dominant arms. The width of the grip was noted during the pre-intervention assessment and kept constant for an individual during the subsequent post-intervention assessment. Muscle strength was recorded as the best (highest) value for the dominant and non-dominant sides as well as average value of the 3 measurements.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
kg
  Dominant hand, At Baseline | 9.7 (3.9) | 9.4 (3.7) | 9.8 (3.4)
  Dominant hand, after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Dominant hand, after 4 months | 11.1 (3.4) | 10.6 (3.0) | 10.9 (3.2)
  Dominant hand, change after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Dominant hand, change after 4 months | 1.41 (2.52) | 1.21 (2.91) | 1.09 (3.15)
  Non-dominant hand, at Baseline | 8.6 (3.5) | 8.6 (3.5) | 8.5 (3.2)
  Non-dominant hand, after 4 months: number analyzed (Participants) | 95 | 95 | 96
  Non-dominant hand, after 4 months | 9.9 (3.4) | 9.47 (3.0) | 9.6 (2.6)
  Non-dominant hand,change after 4 months: number analyzed (Participants) | 95 | 95 | 96
  Non-dominant hand,change after 4 months | 1.34 (2.55) | 0.72 (2.85) | 1.11 (2.44)

6. Secondary Outcome: Change From Baseline in Time to Fatigue After 4 Months
Description: Time to fatigue is defined as the time in seconds taken for the handgrip to fall from maximal value to 50% of the maximal value. Time to fatigue was measured using Jamar hand dynamometer to assess the muscle strength. In this test, participants were required to sustain a maximal contraction until the force dropped to 50% of its maximal value.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
sec
  At Baseline | 12.31 (6.71) | 12.36 (7.66) | 11.13 (9.85)
  After 4 months: number analyzed (Participants) | 95 | 95 | 96
  After 4 months | 14.71 (7.2457) | 14.62 (6.35) | 14.03 (7.25)
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 96
  Change from baseline after 4 months | 2.64 (6.37) | 2.03 (8.39) | 2.78 (6.26)

7. Secondary Outcome: Change From Baseline in Rate of Decline of Muscle Strength After 4 Months
Description: Rate of decline of muscle strength was assessed to measure the muscle endurance of forearm. Sustained isometric contraction of forearm flexors to 50% of maximal handgrip was measured using the Jamar hand dynamometer and was performed on the non-dominant arm. The participant was required to sustain a maximal contraction until the force dropped to 50% of its maximal value. Rate of decline of muscle strength was calculated as 50 percent of maximal value of contraction divided by time to fatigue (50%maximal value of contraction (MVC)/Time to fatigue).
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/sec
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
kg/sec
  At Baseline | 0.38 (0.23) | 0.38 (0.24) | 0.42 (0.26)
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 0.36 (0.17) | 0.33 (0.16) | 0.35 (0.16)
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 96
  Change from baseline after 4 months | -0.01 (0.25) | -0.05 (0.27) | -0.06 (0.28)

8. Secondary Outcome: Change From Baseline in Hemoglobin Level After 4 Months
Description: Hemoglobin level was measured to assess the iron status in study participants.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: gram per decilitre (g/dl)
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
gram per decilitre (g/dl)
  At Baseline | 12.9 [12.3 to 13.4] | 12.94 [12.50 to 13.60] | 12.88 [12.30 to 13.48]
  After 4 months | 12.7 [12.0 to 13.1] | 12.60 [11.80 to 13.30] | 12.60 [12.05 to 13.15]
  Change from baseline after 4 months | -0.20 [-0.70 to 0.20] | -0.31 [-0.80 to 0.10] | -0.20 [-0.70 to 0.10]

9. Secondary Outcome: Change From Baseline in Ferritin Level After 4 Months
Description: Ferritin level was measured to assess the iron status of study participants.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nanogram per mililitre (ng/mL)
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
nanogram per mililitre (ng/mL)
  At Baseline | 27.59 [17.32 to 45.46] | 20.17 [13.14 to 28.96] | 24.48 [16.88 to 39.76]
  After 4 months: number analyzed (Participants) | 93 | 94 | 95
  After 4 months | 38.78 [29.06 to 54.95] | 23.89 [14.58 to 34.34] | 25.79 [16.92 to 36.92]
  Change from baseline after 4 months: number analyzed (Participants) | 92 | 91 | 92
  Change from baseline after 4 months | 9.36 [2.42 to 17.61] | 1.94 [-1.18 to 8.89] | 0.17 [-5.44 to 6.64]

10. Secondary Outcome: Change From Baseline in Soluble Transferring Receptors (sTr) After 4 Months
Description: Soluble transferring receptors (sTr) was measured to assess the iron status of study participants.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: miligram per litre (mg/L)
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
miligram per litre (mg/L)
  At Baseline | 5.91 [5.27 to 7.16] | 6.20 [5.56 to 7.34] | 5.98 [5.29 to 6.94]
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 5.75 [5.11 to 6.65] | 5.99 [5.18 to 7.48] | 6.01 [5.35 to 6.56]
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Change from baseline after 4 months | -0.33 [-0.95 to 0.20] | -0.24 [-0.69 to 0.24] | -0.02 [-0.40 to 0.43]

11. Secondary Outcome: Change From Baseline in C-reactive Protein Level After 4 Months
Description: C-reactive protein level was measured.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
mg/L
  At Baseline | 0.20 [0 to 0.70] | 0.30 [0 to 0.78] | 0.40 [0 to 0.80]
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 0.40 [0 to 0.80] | 0.20 [0 to 0.80] | 0.40 [0.10 to 0.70]
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Change from baseline after 4 months | 0 [-0.20 to 0.40] | 0 [-0.50 to 0.30] | 0 [-0.40 to 0.30]

12. Secondary Outcome: Change From Baseline in Vitamin B2 Level After 4 Months
Description: Vitamin B2 level was measured by erythrocyte glutathione reductase coefficient (EGRAC) method as micronutrient markers in study participants.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
ratio
  At Baseline | 1.56 [1.47 to 1.64] | 1.52 [1.43 to 1.61] | 1.57 [1.48 to 1.70]
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 1.22 [1.17 to 1.28] | 1.47 [1.41 to 1.56] | 1.56 [1.47 to 1.69]
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Change from baseline after 4 months | -0.32 [-0.41 to -0.26] | -0.04 [-0.10 to 0.00] | 0.00 [-0.08 to 0.07]

13. Secondary Outcome: Change From Baseline in Vitamin B6 Level After 4 Months
Description: Vitamin B6 level was measured as micronutrient markers in study participants.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nano mole per litre (nmol/L)
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
nano mole per litre (nmol/L)
  At Baseline: number analyzed (Participants) | 97 | 96 | 98
  At Baseline | 33.77 [20.71 to 50.30] | 34.28 [22.44 to 50.66] | 39.27 [21.76 to 51.98]
  After 4 months: number analyzed (Participants) | 94 | 94 | 96
  After 4 months | 59.66 [39.62 to 79.15] | 37.79 [27.02 to 50.14] | 39.77 [24.29 to 61.77]
  Change from baseline after 4 months: number analyzed (Participants) | 91 | 90 | 95
  Change from baseline after 4 months | 23.96 [6.74 to 45.00] | 4.72 [-5.36 to 16.14] | 2.52 [-11.02 to 19.60]

14. Secondary Outcome: Change From Baseline in Vitamin B12 Level After 4 Months
Description: Vitamin B12 was measured by electrochemilumenesence method as micronutrient markers in study participants.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: picomole per litre(pmol/L)
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
picomole per litre(pmol/L)
  At Baseline | 210.03 [166.77 to 285.74] | 213.02 [163.21 to 296.66] | 224.02 [164.41 to 270.24]
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 427.82 [348.71 to 565.46] | 218.30 [171.22 to 315.05] | 220.44 [158.56 to 272.99]
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Change from baseline after 4 months | 210.77 [164.64 to 266.12] | 5.31 [-25.90 to 28.86] | -10.11 [-39.37 to 15.35]

15. Secondary Outcome: Change From Baseline in Folate Level After 4 Months
Description: Folate level was measured as micronutrient markers in study participants.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nanogram per mililitre (ng/mL)
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
nanogram per mililitre (ng/mL)
  At Baseline | 583.68 [532.68 to 669.43] | 585.29 [543.79 to 644.00] | 592.82 [510.63 to 684.32]
  After 4 months: number analyzed (Participants) | 95 | 95 | 97
  After 4 months | 1013.40 [878.96 to 1147.08] | 592.41 [533.26 to 647.71] | 592.93 [510.63 to 688.04]
  Change from baseline after 4 months: number analyzed (Participants) | 95 | 95 | 97
  Change from baseline after 4 months | 396.97 [286.74 to 496.87] | -13.03 [-49.56 to 40.02] | -9.62 [-56.45 to 48.42]

16. Secondary Outcome: Change From Baseline in Vitamin C Level After 4 Months
Description: Vitamin C level was measured as micronutrient markers in study participants.
Time Frame: Baseline, after 4 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: miligram per decilitre (mg/dL)
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
Number analyzed (Participants) | 100 | 100 | 100
miligram per decilitre (mg/dL)
  At Baseline: number analyzed (Participants) | 96 | 100 | 96
  At Baseline | 0.69 [0.43 to 1.04] | 0.61 [0.41 to 0.98] | 0.72 [0.45 to 1.23]
  After 4 months: number analyzed (Participants) | 95 | 93 | 96
  After 4 months | 1.49 [1.20 to 1.75] | 0.77 [0.46 to 1.19] | 0.76 [0.43 to 1.21]
  Change from baseline after 4 months: number analyzed (Participants) | 92 | 93 | 93
  Change from baseline after 4 months | 0.83 [0.48 to 1.09] | 0.13 [-0.33 to 0.45] | 0.09 [-0.46 to 0.44]

ADVERSE EVENTS:
Description: General Disorders adverse events (AEs) terms are not coded.
Arm/Group | Experimental Group (Fortified Nutritional Supplement) | Control Group A (Unfortified Nutritional Powder) | Control Group B (No Intervention)
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 29/100 | 25/100 | 8/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (Fortified Nutritional Supplement) (N=100) | Control Group A (Unfortified Nutritional Powder) (N=100) | Control Group B (No Intervention) (N=100)
Vomiting (General disorders) | 5 | 2 | 0
Loose stools (General disorders) | 1 | 0 | 0
Skin allergy (General disorders) | 1 | 2 | 0
Abdominal pain (General disorders) | 1 | 0 | 1
Excessive tiredness after 20m shuttle (General disorders) | 1 | 1 | 1
Abrasion during 20 m shuttle (General disorders) | 0 | 1 | 1
Felt dizzy after blood collection (General disorders) | 2 | 1 | 0
Fever (General disorders) | 14 | 8 | 3
Otitis media (General disorders) | 1 | 0 | 0
Urinary tract infection (General disorders) | 0 | 1 | 0
Abrasion (General disorders) | 0 | 1 | 0
Fall/Fracture (General disorders) | 1 | 1 | 1
Chicken pox (General disorders) | 0 | 1 | 0
Leg wound (General disorders) | 1 | 1 | 0
Scabies (General disorders) | 0 | 0 | 1
Tooth ache (General disorders) | 0 | 2 | 0
Respiratory tract infection (General disorders) | 0 | 1 | 0
Ear/leg pain (General disorders) | 0 | 1 | 0
Perianal abscess (General disorders) | 0 | 1 | 0
Insect bite (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.